CLINICAL TRIAL: NCT01374581
Title: A Randomized Clinical Trial to Measure the Impact of Retreatment With an Artemisinin-based Combination on Malaria Incidence and Its Potential Selection of Resistant Strains
Brief Title: Impact of Artemisinin-based Combination Therapy and Quinine on Treatment Failure and Resistance in Uncomplicated Malaria
Acronym: QuinAct
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Fund for Scientific Research, Flanders, Belgium (Other); Institute of Tropical Medicine, Belgium (Other); University of Kinshasa (Other); Centre Muraz (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Jean-Pierre Van geertruyden, Prof, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UA-IHU-2010-01 version 1
Record Dates: First submitted 2011-06-09; First posted 2011-06-16 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Malaria
Keywords: retreatment; artemisinin-based combination; malaria; resistant
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination; Quinine; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artemether/Lumefantrine (Experimental): Tablets 20 mg/120 of Artemether/Lumefantrine will be given to 124 trial patients
  Interventions: Drug: Artemether/Lumefantrine
- Artesunate/Amodiaquine (Experimental): Tablets 25mg/67,5 mg of Artesunate/Amodiaquine will be given to 124 trial patients.
  Interventions: Drug: Artesunate/Amodiaquine
- Quinine + Clindamycin (Active Comparator): Quinine tablet 125mg + Clindamycin syrup 75mg/5ml will be given to 60 children.
  Interventions: Drug: Quinine + Clindamycin

INTERVENTIONS:
Drug: Artemether/Lumefantrine — Tablets containing 20 mg of Artemether and 120 mg of Lumefantrine. Each dose to be taken with high-fat food or drinks (for example milk).
  Weight in kg Number of tablet per dose Age 5 to < 15 kg 1 tablet per dose 15 to < 25 kg 2 tablets per dose 25 to < 35 kg 3 tablets per dose
  Other Names: Coartem®
  Arms: Artemether/Lumefantrine
Drug: Artesunate/Amodiaquine — Age (Weight in Kg) Dose Treatment duration 2 to 11 months (= 4,5 to < 9kg):1 tablet (25 mg/675mg) for 3 days
  1 to 5 years (= 9 kg to < 18 kg)1 tablet(25mg/67,5mg)for 3 days
  Other Names: Co-arsucam®
  Arms: Artesunate/Amodiaquine
Drug: Quinine + Clindamycin — this arm consist to 7 days treatment of 60 patients with quinine tablet 125mg + clindamycin syrup as follow;
  Quinine:
  9 to < 11 kg: ½ tablets 12 to < 19 kg: 1 tablets per dose 20 to < 27 kg: 1½ tablets per dose 28 to < 35 kg: 2 tablets per dose
  Clindamycin syrup:
  10 mg/kg twice daily
  Other Names: Quinimax® tablet 125mg; Dalacin® syrup 75mg/5ml
  Arms: Quinine + Clindamycin

SUMMARY:
This is a bi-centric phase IIIb, randomized, open label, 3-arm clinical trial performed to investigate the impact of retreatment with an Artemisinin-Based Combination (ACT), for example Arthemeter-Lumefantrine (AL) in Uganda (Ug) and artesunate-amodiaquine (ASAQ) in RDCongo, on malaria incidence and its potential selection of resistant strains.

Patients will be followed-up for efficacy and safety during 42 days after treatment with the first line therapy recommended by the national authorities(arthemeter-lumefantrine in Uganda and artesunate-amodiaquine in RDCongo) and retreated the patients either with the same ACT or an other ACT or oral Quinine + clyndamicin.

The investigators hypothesize that (re)treatment with the first line ACT treatment beyond 14 days is as efficacious as any other rescue treatment, without the risk of selecting drug resistant strains.

DETAILED DESCRIPTION:
RATIONALE Following the World Health Organization (WHO) guidelines, most African countries have opted for ACT. Several clinical trials on ASAQ, an ACT, completed in Africa have shown an efficacy > 90% (3-5). Furthermore, after The polymerase chain reaction (PCR) analysis, over 75 % of ASAQ & AL treatment failures have been classified as new infections, while recrudescences have low parasite densities. ASAQ is safe and easy administered, with a good treatment adherence. Therefore, effectiveness may be close to efficacy . ASAQ has now been developed as fixed-dose combination and registered. The Democratic Republic of Congo (DRC) has also chosen ASAQ as first-line treatment for uncomplicated malaria.

Efficacy of the 6 dose regimen of AL has been demonstrated in semi-immune and non-immune populations in Asia and Africa to be consistently greater than 95%, with rapid parasite and symptom clearance and significant gametocidal effect. In Uganda, AL has already been chosen as first-line treatment for uncomplicated malaria.

In DRC and Uganda, quinine is the rescue treatment for malaria. It is cheap, widely available and generally considered to be effective but is not popular due to the unwanted side effects. Quinine has a very short half life, therefore repeated dosing is required. In an efficacy study of quinine and artemisinin for uncomplicated malaria in Vietnam, recrudescence rates were 16% after 7 days of quinine monotherapy. In studies conducted in Gabon, Plasmodium falciparum in Vitro sensitivity to quinine was high and had not changed over the past decade. Although quinine monotherapy shows high efficacy in the setting of clinical trials, it has considerable disadvantages, mainly because of its poor tolerability and the prolonged treatment course. Poor adherence carries a high risk of treatment failure, particularly because quinine causes a syndrome of adverse effects known as cinchonism that includes primarily tinnitus, nausea, and vertigo. Other reported side effects are high tone hearing impairment, dizziness, hypotension as well as headache and visual disturbances. As result of these side effects, some studies have reported poor compliance to treatment. A randomized trial in Thailand reported 71% adherence Such poor adherence to the 7-days regimen is associated with a high risk of treatment failure, which can contribute to the development and spread of resistance. Furthermore, in field circumstances patients are often re-treated with the recommended first line drug, i.e. ASAQ.

As quinine is effective against all species of malaria including chloroquine-resistant strains of P. falciparum, it is widely used for the treatment of severe malaria. Therefore, it should be protected from resistance by a rational use, as its effectiveness in uncomplicated malaria is lower than ACT.

Rationale Considering the facts that: over 90% of treatment failure to ASAQ or AL are new infections, parasitaemia is low in case of recrudescence occurring from day 14 and in real-life situations patients are re-treated with the same first line drug, there is the need to assess the role of the first line treatment as rescue treatments. This efficacy will be compared to quinine + clindamycin and another ACT treatment in line with the WHO guideline, and another ACT treatment to provide clear guidelines. The investigators hypothesize that re-treatment with the first line ACT treatment beyond 14 days is as efficacious as any other rescue treatment, without the risk of selecting drug resistant strains. Furthermore, a prolonged follow up will allow the assessment of the epidemiological, parasite related risk factors for repeated malaria infection and to collect samples for immunological risk factors for repeated malaria attacks.

TRIAL OBJECTIVES AND PURPOSE

Efficacy

The primary objective is:

1. to show that, in children aged 12 to 59 months with recurrent uncomplicated P. falciparum malaria within 42 days of treatment with an artemisinin-based combination therapy (ASAQ in DRC or AL in Uganda), the PCR adjusted efficacy at 28 days after re-treatment with the same artemisinin-based combination therapy is at least 90% and
2. to estimate the relative efficacy of re-treatment with the same artemisinin-based combination compared to treatment with quinine and treatment with another artemisinin-based combination therapy (ASAQ after first line AL treatment or AL after first line ASAQ treatment).

Secondary objectives are:

1. To evaluate the PCR-unadjusted efficacy at 28 days of re-treatment with the same artemisinin-based combination therapy and to compare it to treatment with quinine + clindamycin and treatment with another artemisinin-based combination therapy (ASAQ after first line AL treatment or AL after first line ASAQ treatment).
2. To evaluate and compare the efficacy of AL, ASAQ and quinine + clindamycin as rescue treatment for a recurrent P. falciparum malaria episode occurring 2 weeks after the administration of the first line treatment, with and without PCR adjustment.
3. To evaluate and compare the 42 days clinical efficacy of AL (Uganda) and ASAQ (RDC) for the first line treatment of uncomplicated P. falciparum malaria, with and without PCR adjustment.
4. To evaluate and compare the efficacy of the different rescue treatment regimens in terms of fever clearance time, asexual parasite clearance time, gametocytaemia at day 7, 14, 21 and 28, and, Hemoglobin changes between day 0 and days 14 and 28.

Additional objectives are:

1. To evaluate the selection of Plasmodium falciparum pfmdr1 alleles following therapy with quinine + clindamycin, AL and ASAQ.
2. To assess epidemiological, parasitological and host related predictors for recurrent malaria infections, an adjacent study that will be developed in a separate nested study protocol.

Safety To evaluate the safety and tolerability of AL, ASAQ and quinine + clindamycin when used as rescue treatments.

DRUG TO BE TESTED Quinine Quinamax® (Sanofi) + Clindamycin Dalacin® (Pfizer): in this study the investigators will use Dalacin syrup (75mg/5ml) and dry Quinamax® tablets (125mg) of whom the dosage is not adapted to children below 9 kg. The latter explains why children below 12 months will be exclude from our study

Artemether-lumefantrine (AL) AL of Novartis, marketed under the trademarks Riamet® and Coartem®, was registered in Switzerland in 1999, it is pre-qualified by the WHO and has since received marketing authorisation in several endemic and non-endemic countries. A recent review showed that the drug combination is highly efficacious against sensitive and multidrug resistant falciparum malaria as it offers the advantage of rapid clearance of parasites by artemether and the slower elimination of residual parasites by lumefantrine.

Amodiaquine artesunate ASAQ is safe, easy to use and efficacious and the second most used ACT worldwide. DRC, through the National Malaria Control Program has complied with the WHO recommendation by recommending since 2005 ASAQ as first line treatment for uncomplicated malaria. In a study conducted in 2004 in the eastern part of the country, the efficacy of ASAQ was estimated at 93% after PCR adjustment. Twenty five trials (11,700 patients) carried out in Sub-Saharan Africa show a PCR-adjusted efficacy at day 28 of 94%. ASAQ is currently the second most used ACT globally (co formulated Co-arsucam® or ASAQ Winthrop®, Sanofi-Aventis. A study has been conducted in Burkina Faso in children under 5 and has shown that co-formulated ASAQ is well tolerated and its efficacy was 93% after PCR correction. The investigators will use this co-formulated ASAQ Winthrop® of Sanofi-Aventis, age dosed and put on the market since March 2007. This product has been pre-qualified by the WHO.

STUDY DESIGN This is a bi-centre, phase IIIb, randomized, open label, 3-arm trial.

ELIGIBILITY:
Inclusion Criteria:

1. Have been enrolled in the first phase
2. Recurrent Plasmodium falciparum infection with clinical symptoms.
3. Parents' or guardians' willingness and ability to comply with the study protocol for the duration of the study.
4. Signed (or thumb-printed whenever parents/guardians are illiterate) (second) informed consent by the parents or guardians. Note: the informed consent will cover the whole period of the study, including additional active follow ups

Exclusion Criteria:

Patients with at least one of the following criteria will be excluded:

1. Participation in any other investigational drug study (antimalarial or others) during the previous 30 days.
2. Known hypersensitivity and previous Serious Adverse Events related to the study drugsto the study drugs.
3. Severe malaria( WHO 2000) or danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand.
4. Presence of intercurrent illness or any condition (cardiac, renal, hematologic, hepatic diseases) which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study, including known G6PD deficiency.
5. Patients who are taking drug which may prolong the QT (imidazole and triazole, antifungal agent).
6. Severe malnutrition (defined as weight for height <70% of the median NCHS/WHO reference).
7. Ongoing prophylaxis with drugs having antimalarial activity such as cotrimoxazole for the prevention of Pneumocisti carini pneumonia in children born to HIV+ women.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2117 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Late Parasitological Failure | Day4-Day28
  Parasitaemia after day 3 in the absence of fever (axillary temperature <37.5°C)

SECONDARY OUTCOMES:
PCR unadjusted efficacy | Day 28 days
  Proportion of children without (PCR not adjusted) treatment failure (TF28U): all treatment failures detected during the active follow up, regardless of genotyping.
Day 42 clinical efficacy | Day 42
  All clinical treatment failures detected during the 42 days follow up for the first line treatment, with and without PCR adjustment. As no active monitoring of parasitaemia after day 3 is planned this includes ETF and LCF following WHO criteria.
Change in Fever clearance time (FCT) | Day 0, Day 1, Day 2
  The time (in days) from the time of randomization to the first two consecutive measurements on 2 different days of axillary temperature below 37.5°C.
Change in Asexual parasite clearance time | Day 0, Day 1, Day 2
  Asexual parasite clearance time is defined as the time (in days) from time of randomization to 2 consecutive negative blood slides (collected at different days). The time to the event will be taken as the time to the first negative slide.
  5. Gametocytaemia (prevalence and density) at day 7, 14, 21 and 28 after treatment.
Hb changes | Day 0, Days 14 and Day 28
  Variation in Hb level between two measurements.
Early Treatment Failure | Day0-Day3
  Development of danger signs or severe malaria on Day 0, Day 1 Day 2 or Day 3, in the presence of parasitaemia Parasite density on Day 2 > Day 0 count, irrespective of axillary temperature Presence of parasitaemia on Day 3 with fever (axillary temperature ≥ 37.5°C) Parasitaemia on Day 3 ≥ 25 % of count on Day 0.
Late Clincial Failure | Day0-Day28
  Development of danger signs or severe malaria after Day 3 in the presence of parasitaemia Presence of parasitaemia and fever on any day from Day 4 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Hypolite M. Mavoko, MD MPH, Principal Investigator — Kinshasa University, RDCongo; Carolyn Nabasumba, M.B.Ch.B, Principal Investigator — Kazo health centre IV Uganda; Jean-Pierre Van geertruyden, MD MPH PhD, Study Director — International Health Unit Antwerp university
Locations (2):
- Centre de Santé Lisungi, Kinshasa, Mont-Ngafula, Republic of the Congo
- Kazo Health centre IV, Kiruhura, Uganda

REFERENCES:
- [Derived] Mavoko HM, Nabasumba C, da Luz RI, Tinto H, D'Alessandro U, Kambugu A, Baraka V, Rosanas-Urgell A, Lutumba P, Van Geertruyden JP. Efficacy and safety of re-treatment with the same artemisinin-based combination treatment (ACT) compared with an alternative ACT and quinine plus clindamycin after failure of first-line recommended ACT (QUINACT): a bicentre, open-label, phase 3, randomised controlled trial. Lancet Glob Health. 2017 Jan;5(1):e60-e68. doi: 10.1016/S2214-109X(16)30236-4. Epub 2016 Nov 11. PMID 27840069
- [Derived] Muhindo Mavoko H, Kalabuanga M, Delgado-Ratto C, Maketa V, Mukele R, Fungula B, Inocencio da Luz R, Rosanas-Urgell A, Lutumba P, Van Geertruyden JP. Uncomplicated Clinical Malaria Features, the Efficacy of Artesunate-Amodiaquine and Their Relation with Multiplicity of Infection in the Democratic Republic of Congo. PLoS One. 2016 Jun 9;11(6):e0157074. doi: 10.1371/journal.pone.0157074. eCollection 2016. PMID 27280792
- [Derived] Muhindo Mavoko H, Nabasumba C, Tinto H, D'Alessandro U, Grobusch MP, Lutumba P, Van Geertruyden JP. Impact of retreatment with an artemisinin-based combination on malaria incidence and its potential selection of resistant strains: study protocol for a randomized controlled clinical trial. Trials. 2013 Sep 23;14:307. doi: 10.1186/1745-6215-14-307. PMID 24059911